CLINICAL TRIAL: NCT02357472
Title: The Effect of a Higher Dose of Dehydroepiandrosterone (DHEA) Supplementation on the Number of Oocytes Obtained During IVF in Poor Ovarian Responders
Brief Title: The Effect of a Higher Dose of Dehydroepiandrosterone (DHEA) Supplementation in Poor Responders
Acronym: DHEA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Many patients couldn't wait for DHEA treatment for three months.
Sponsor: ShangHai Ji Ai Genetics & IVF Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: JIAIE2014-03
Record Dates: First submitted 2015-01-17; First posted 2015-02-06 (Estimated); Results first posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Infertility
Keywords: Reproductive aging; DHEA; poor ovarian responder
MeSH Terms: conditions — Infertility | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High dose group (Experimental): dehydroepiandrosterone,DHEA,capsule, 50mg/capsule, one capsule t.i.d..
  Interventions: Dietary Supplement: dehydroepiandrosterone
- Standard dose group (Other): dehydroepiandrosterone,DHEA, capsule, 25mg/capsule, one capsule t.i.d.
  Interventions: Dietary Supplement: dehydroepiandrosterone

INTERVENTIONS:
Dietary Supplement: dehydroepiandrosterone — high dose group treatment represent for 50mg t.i.d. Patients in these group will take one capsule each time and three times a day for three months before entering into IVF cycles.
  Other Names: DHEA (Lab Hercules™)

SUMMARY:
The supplementation of Dehydroepiandrosterone (DHEA) has been used in some centers for patients with previous poor ovarian reserve and response in an attempt to improve pregnancy outcomes. However, there still has controversy on the clinical effect on the 75mg/d for the use,especially in Asian people. Whether the double dosage of DHEA in patients with poor ovarian reserve and response in China can improve the IVF outcome with little side effect is unknown.

The aim of this randomized controlled study is to compare the effect of a higher dose (150mg daily) and a standard dose (75mg daily) of DHEA on the number of oocytes obtained in poor ovarian responders. The effect of DHEA action on the cumulus cells will be examined.

DETAILED DESCRIPTION:
Consecutive infertile women attending the subfertility clinic at Shang Hai Ji Ai Genetics &IVF Institute for IVF treatment will be approached. Those fulfilling the selection criteria stated below would be recruited and a written consent will be obtained after detailed explanation and counseling.

Poor ovarian responders are defined according to the Bologna criteria fulfilling 2 out of 3 of the following:

(i) Advanced maternal age (>/= 40) or any other genetic or acquired risk factor for poor ovarian response(POR); (ii) Previous poor ovarian response (POR) (</= 3 oocytes with a conventional stimulation protocol using at least 150 international units (IU) gonadotrophins per day) (iii) Abnormal ovarian reserve test [i.e. antral follicle count (AFC) < 5-7 or antimüllerian hormone (AMH) < 0.5 - 1.1ng/ml]

Alternatively, two episodes of POR after maximal stimulation are sufficient to define a patient as poor responder in the absence of advanced maternal age or abnormal ovarian reserve test(ORT).

Baseline assessment will be performed at early follicular phase (Day 2 or 3) at recruitment. Patient characteristics including age, Body Mass Index (BMI), and smoking status would be recorded and blood test including follicular stimulating hormone (FSH), estradiol (E2), testosterone, DHEA-S, full blood count, renal and liver function test would be checked. Pelvic scan will be performed to assess the total AFC and total ovarian volume.

Subjects will be randomized divided into two groups:

1. Standard dose group: Subjects will take DHEA (Lab Hercules™) 25mg three times a day for 12 weeks prior to the start of IVF treatment till the day of egg collection.
2. High dose group: Subjects will taking DHEA (Lab Hercules™) 50mg three times a day for 12 weeks prior to the start of IVF treatment till the day of egg collection.

Hormonal profile, ultrasound assessment, full blood count, renal and liver function test will be repeated in follicular phase (D2 or 3) of every month or cycle followed by a IVF treatment using antagonist protocol based on our standard departmental regimen. The human menopausal gonadotropin (hMG) injections were started at 300 international units (IU) for 2 days followed by 300 international units (IU) daily. Improvement of ovarian reserve markers would be assessed by the change in serum AMH between the time of recruitment and that after 6 and 12 weeks of DHEA. Cycle characteristics including the dose of gonadotrophins use, duration of stimulation, number of oocytes obtained, number of fertilized embryos and good quality embryos will be recorded and follicular fluid will be saved for hormonal profiles.

Statistics

1. Statistical tests

   Statistical comparisons will be performed according to the intention to treat principle by Student t test or Fisher's exact tests for normally distributed data and Mann-Whitney test for skewed data. Chi-square test would be used for binary variables. Statistical analyses will be performed using the Statistical Package for (the) Social Sciences (SPSS) software and a P-value of 0.05 would be considered statistically significant. Linear regression analysis / logistic regression analysis curve would be used to evaluate the age, BMI, smoking, FSH, E2, AMH, testosterone, DHEA-S, AFC, ovarian volume and duration of DHEA use for the prediction of improved ovarian reserve after DHEA supplementation.
2. Sample size estimation

The number of oocytes retrieved will be used as the primary outcome of the study. Based on our own database for patients undergoing IVF treatment, the mean oocytes obtained was 2.7 with a standard deviation (SD) of 1.4. Assuming an increase of oocytes obtained by 1.0 to be clinically significant, 18 subjects in each arm would be required to achieve a test of significance of 0.05 and a power of 0.8. Considering possible dropouts, we aim at recruiting 18 patients in each arm, i.e. 36 patients.

In order to compare one of the secondary outcome -- AMH (which has more relevance on the effect of ovarian response) with adequate power, based on our own database for patients undergoing IVF treatment, the mean AMH of the group with poor ovarian reserve is 0.8 with a SD of 0.6. Assuming an increase of number of oocyte retrieved by 0.5 to be clinically significant, 25 subjects in each arm would be required to achieve a test of significance of 0.01 and a power of 0.9. Totally 50 patients.

ELIGIBILITY:
Inclusion Criteria:

1. age<45 years,
2. subfertility >1 year, and
3. A previous POR (≤3 oocytes with a conventional stimulation protocol of at least 150 IU FSH per day); or
4. An abnormal ovarian reserve test (i.e. AFC ≤5-7 follicles or AMH ≤0.5-1.1 ng/ml).

Exclusion Criteria:

Patients were excluded if they:

1. had a history of ovarian cystectomy or oophorectomy,
2. had received cytotoxic chemotherapy,
3. had received pelvic irradiation, or
4. had a history of taking testosterone or DHEA supplementation

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2015-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Xi Sun, PHD,MD, Study Chair — Shang Hai JIAi genetics & IVF center; Jing Fu, MD, Principal Investigator — Shang Hai JIAi genetics & IVF center; Ying Su Liu, PHD,MD, Study Director — Shang Hai JIAi Genetics & IVF center
Locations (1):
- Ji Ai Genetics and IVF center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jenkins JM, Davies DW, Devonport H, Anthony FW, Gadd SC, Watson RH, Masson GM. Comparison of 'poor' responders with 'good' responders using a standard buserelin/human menopausal gonadotrophin regime for in-vitro fertilization. Hum Reprod. 1991 Aug;6(7):918-21. doi: 10.1093/oxfordjournals.humrep.a137459. PMID 1761658
- [Background] Ulug U, Ben-Shlomo I, Turan E, Erden HF, Akman MA, Bahceci M. Conception rates following assisted reproduction in poor responder patients: a retrospective study in 300 consecutive cycles. Reprod Biomed Online. 2003 Jun;6(4):439-43. doi: 10.1016/s1472-6483(10)62164-5. PMID 12831590
- [Background] Keay SD, Liversedge NH, Mathur RS, Jenkins JM. Assisted conception following poor ovarian response to gonadotrophin stimulation. Br J Obstet Gynaecol. 1997 May;104(5):521-7. doi: 10.1111/j.1471-0528.1997.tb11525.x. No abstract available. PMID 9166190
- [Background] Casson PR, Lindsay MS, Pisarska MD, Carson SA, Buster JE. Dehydroepiandrosterone supplementation augments ovarian stimulation in poor responders: a case series. Hum Reprod. 2000 Oct;15(10):2129-32. doi: 10.1093/humrep/15.10.2129. PMID 11006185
- [Background] Barad DH, Gleicher N. Increased oocyte production after treatment with dehydroepiandrosterone. Fertil Steril. 2005 Sep;84(3):756. doi: 10.1016/j.fertnstert.2005.02.049. PMID 16169414
- [Background] Barad D, Gleicher N. Effect of dehydroepiandrosterone on oocyte and embryo yields, embryo grade and cell number in IVF. Hum Reprod. 2006 Nov;21(11):2845-9. doi: 10.1093/humrep/del254. Epub 2006 Sep 22. PMID 16997936
- [Background] Barad D, Brill H, Gleicher N. Update on the use of dehydroepiandrosterone supplementation among women with diminished ovarian function. J Assist Reprod Genet. 2007 Dec;24(12):629-34. doi: 10.1007/s10815-007-9178-x. Epub 2007 Dec 11. PMID 18071895
- [Background] Gleicher N, Ryan E, Weghofer A, Blanco-Mejia S, Barad DH. Miscarriage rates after dehydroepiandrosterone (DHEA) supplementation in women with diminished ovarian reserve: a case control study. Reprod Biol Endocrinol. 2009 Oct 7;7:108. doi: 10.1186/1477-7827-7-108. PMID 19811650
- [Background] Hartkamp A, Geenen R, Godaert GL, Bijl M, Bijlsma JW, Derksen RH. Effects of dehydroepiandrosterone on fatigue and well-being in women with quiescent systemic lupus erythematosus: a randomised controlled trial. Ann Rheum Dis. 2010 Jun;69(6):1144-7. doi: 10.1136/ard.2009.117036. Epub 2009 Oct 22. PMID 19854713
- [Background] Casson PR, Santoro N, Elkind-Hirsch K, Carson SA, Hornsby PJ, Abraham G, Buster JE. Postmenopausal dehydroepiandrosterone administration increases free insulin-like growth factor-I and decreases high-density lipoprotein: a six-month trial. Fertil Steril. 1998 Jul;70(1):107-10. doi: 10.1016/s0015-0282(98)00121-6. PMID 9660430

RESULTS

PARTICIPANT FLOW:
Groups:
- Standard Dose Group: dehydroepiandrosterone,DHEA, capsule, 25mg/capsule, one capsule t.i.d.
  dehydroepiandrosterone: high dose group treatment represent for 50mg t.i.d and standard dose group represents for normal treatment with 25mg t.i.d. Each patients in these two group will take one capsule each time and three times a day for three months before entering into IVF cycles.
- High Dose Group: dehydroepiandrosterone,DHEA,capsule, 50mg/capsule, one capsule t.i.d..
  dehydroepiandrosterone: high dose group treatment represent for 50mg t.i.d and standard dose group represents for normal treatment with 25mg t.i.d. Each patients in these two group will take one capsule each time and three times a day for three months before entering into IVF cycles.
Period: Overall Study
Arm/Group | Standard Dose Group | High Dose Group
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Dose Group | Standard Dose Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 30 | 60
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.40 (4.70) | 37.68 (5.40) | 38.3 (5.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number of Oocytes Obtained
Description: After 12 weeks treatment, the number of oocytes obtained will be detected from the higher dose group and standard dose group
Time Frame: After taking DHEA for 12 weeks
Measure: Mean (Standard Error); unit: oocytes
Arm/Group | High Dose Group | Standard Dose Group
Number analyzed (Participants) | 30 | 30
oocytes | 3.82 (0.28) | 2.51 (0.22)
Statistical Analysis 1: Comparison: High Dose Group vs Standard Dose Group; It was caculated that 60 paticipants randomized in a 1:1between 2 arms would would have at least 85% power to detect a difference of 1.32 oocytes between the high dose group and standard dose group after 12 weeks.Sample size was determined using 2 sided 2 sample t-test (α = 0.05).Assumptions included a common standard deviation of 1.72; Test type: Non-Inferiority or Equivalence — Sample Size to Achieve 0.80 Power to Test Equivalency at the α = 0.05 Significance Level for True Proportions; p = 0.0003, t-test, 2 sided; Mean Difference (Final Values) = 1.31, 95% CI 2-sided [0.6216 to 2.002], Standard Error of Mean 1.31

2. Secondary Outcome: AFC
Description: Antral follicle count (AFC)
Time Frame: After taking DHEA for 12 weeks
Population: The patients who took DHEA for 12 weeks
Measure: Mean (Standard Error); unit: follicles
Groups:
- High Dose Group: The patients who took 50mg t.i.d. DHEA for 12 weeks
- Standard Dose Group: The patients who took DHEA 25mg t.i.d.for 12 weeks
Arm/Group | High Dose Group | Standard Dose Group
Number analyzed (Participants) | 30 | 30
follicles | 4.00 (0.20) | 4.66 (0.26)

3. Secondary Outcome: Follicle Stimulating Hormone (FSH) Levels
Description: The change of FSH levels in the three groups.
Time Frame: 12 weeks after taking DHEA
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | High Dose Group | Standard Dose Group
Number analyzed (Participants) | 30 | 30
IU/L | 12.84 (0.99) | 11.69 (0.83)

4. Secondary Outcome: E2
Description: Serum E2 levels
Time Frame: 12 weeks after taking DHEA
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | High Dose Group | Standard Dose Group
Number analyzed (Participants) | 30 | 30
pmol/L | 51.88 (5.64) | 39.11 (4.44)

5. Secondary Outcome: The Number of Follicles>10mm
Description: The number of follicles>10mm represent for the ovarian reserve and response
Time Frame: 12 weeks after taking DHEA
Measure: Mean (Standard Deviation); unit: follicles
Arm/Group | High Dose Group | Standard Dose Group
Number analyzed (Participants) | 30 | 30
follicles | 8.24 (0.32) | 3.71 (0.24)

6. Secondary Outcome: AMH
Description: The change of AMH levels in serum
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- High Dose Group: The patients have taken DHEA 50mg t.i.d.for 12 weeks when they came to enter the IVF cycle.
- Standard Dose Group: The patients have taken DHEA 25mg t.i.d.for 12weeks when they came to enter the IVF cycle.
Arm/Group | High Dose Group | Standard Dose Group
Number analyzed (Participants) | 30 | 30
ng/ml | 3.05 (0.42) | 1.62 (0.15)

7. Secondary Outcome: Testosterone
Time Frame: 12 weeks after taking DHEA
Measure: Mean (Standard Deviation); unit: ng/dl
Groups:
- High Dose Group: The patients took DHEA 50mg t.i.d. for 12 weeks.
- Standard Dose Group: The patients took DHEA 25mg t.i.d. for 12weeks.
Arm/Group | High Dose Group | Standard Dose Group
Number analyzed (Participants) | 30 | 30
ng/dl | 31.67 (2.6) | 31.59 (1.94)

8. Secondary Outcome: Dehydroepiandrosterone-Sulfide (DHEA-S)
Time Frame: 12 weeks after taking DHEA
Measure: Mean (Standard Deviation); unit: ug/ml
Arm/Group | High Dose Group | Standard Dose Group
Number analyzed (Participants) | 30 | 30
ug/ml | 2.69 (0.24) | 1.75 (0.20)

9. Secondary Outcome: Insulin-like Growth Factor-1 (IGF-1)
Time Frame: 12 weeks after taking DHEA
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | High Dose Group | Standard Dose Group
Number analyzed (Participants) | 30 | 30
ng/ml | 90.87 (6.50) | 71.85 (4.39)

10. Other Pre Specified Outcome: The Number of Mature Oocytes Obtained
Time Frame: up to 12 weeks
Measure: Mean (Standard Deviation); unit: oocytes
Arm/Group | High Dose Group | Standard Dose Group
Number analyzed (Participants) | 30 | 30
oocytes | 4.1 (0.24) | 1.93 (0.27)

11. Other Pre Specified Outcome: Pregnancy Rate
Description: The rate of clinical pregnancy
Time Frame: 2 weeks after transfer
Measure: Number; unit: percentage of pregnancy
Arm/Group | High Dose Group | Standard Dose Group
Number analyzed (Participants) | 30 | 30
percentage of pregnancy | 7 | 4

12. Other Pre Specified Outcome: the Numbers of Fertilized Embryos
Time Frame: 12 weeks after taking DHEA
Measure: Mean (Standard Deviation); unit: embryos
Arm/Group | High Dose Group | Standard Dose Group
Number analyzed (Participants) | 30 | 30
embryos | 1.70 (0.17) | 1.92 (0.21)

13. Other Pre Specified Outcome: the Numbers of Cleaved Embryos
Time Frame: After taking DHEA for 12 weeks
Measure: Mean (Standard Deviation); unit: embryos
Arm/Group | High Dose Group | Standard Dose Group
Number analyzed (Participants) | 30 | 30
embryos | 1.63 (0.19) | 1.89 (0.23)

14. Other Pre Specified Outcome: the Numbers of Top-quality Embryos.
Description: top-quality embryos are represented for >7cell on Day 3 and the fragments <20%
Time Frame: 12 weeks after taking DHEA
Measure: Mean (Standard Deviation); unit: embryos
Arm/Group | High Dose Group | Standard Dose Group
Number analyzed (Participants) | 30 | 30
embryos | 1.11 (0.15) | 0.85 (0.13)

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- High Dose Group: The patients took DHEA 50mg t.i.d. for three months before entering into IVF cycles.
- Standard Dose Group: The patients took DHEA 25mg t.i.d. for three months before entering into IVF cycles.
Arm/Group | High Dose Group | Standard Dose Group
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
The primary outcome measure is oocyte obtained not the IVF clinical pregnancy and the early termination leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No